CLINICAL TRIAL: NCT00870454
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled Study of Carisbamate in the Treatment of Neuropathic Pain in Diabetic Peripheral Neuropathy Followed by a Blinded Extension Phase
Brief Title: An Efficacy and Safety Study of Carisbamate in the Treatment of Nerve Pain in Diabetics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR015973; CARISNPP2003
Record Dates: First submitted 2009-03-25; First posted 2009-03-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Diabetic Neuropathies
Keywords: Diabetic neuropathies; Diabetic neuropathy, painful; Carisbamate; Neurotherapeutic agents
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Pregabalin; S-2-O-carbamoyl-1-o-chlorophenyl-ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 001 (Experimental): Carisbamate 800 mg/d 200 mg/d twice daily titrated up to 400 mg twice daily as tolerated by Week 3
  Interventions: Drug: Carisbamate 800 mg/d
- 002 (Experimental): Carisbamate 1 200 mg/d 200 mg/d twice daily titrated up to 600 mg twice daily as tolerated by Week 3
  Interventions: Drug: Carisbamate 1,200 mg/d
- 003 (Active Comparator): Pregabalin 300 mg/d 75 mg/d twice daily for Week 1 followed by 150 mg twice daily for the remainder
  Interventions: Drug: Pregabalin 300 mg/d
- 004 (Placebo Comparator): Placebo Placebo capsules twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin 300 mg/d — 75 mg/d twice daily for Week 1, followed by 150 mg twice daily for the remainder
  Arms: 003
Drug: Carisbamate 800 mg/d — 200 mg/d twice daily, titrated up to 400 mg twice daily, as tolerated, by Week 3
  Arms: 001
Drug: Carisbamate 1,200 mg/d — 200 mg/d twice daily, titrated up to 600 mg twice daily, as tolerated, by Week 3
  Arms: 002
Drug: Placebo — Placebo capsules twice daily
  Arms: 004

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of carisbamate (800 and 1200 mg/day) in patients with diabetic neuropathic pain.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned by chance), double-blind (neither the investigator or the patient knows the name of the study assigned drug), placebo- and active-controlled, parallel-group, multicenter study, with an optional extension phase, in patients with diabetic peripheral neuropathy (DPN), or nerve pain in their lower extremities resulting from diabetes. The study population includes men and women between 18 and 75 years of age who have chronic neuropathic pain associated with diabetic neuropathy. Up to 440 subjects will be enrolled and randomly assigned (like flipping a coin) in a 1:1:1:1 ratio to treatment with carisbamate 800 milligrams per day (mg/d), carisbamate 1,200 mg/d, pregabalin 300 mg/d, or placebo. The double-blind treatment will be administered orally, in a twice-daily regimen, with or without food, over a period of 15 weeks. The study will consist of a pretreatment phase, including a screening, washout, and baseline period; a double-blind treatment phase, with a titration and a fixed-dosage period; an optional blinded extension phase (with carisbamate 400 to 1,200 mg/d or pregabalin 150 to 300 mg/d); and a posttreatment phase (including a follow-up visit and telephone contact). The duration of the study (excluding the pretreatment phase) is approximately 58 weeks for patients who decide to enter the extension phase and approximately 19 weeks for the other patients. The pretreatment phase will last up to 28 days, including a screening visit up to 28 days before the planned first dose of study drug, a washout of up to 7 days for subjects who need to discontinue medications, and a baseline period of at least 7 days to determine daily average DPN scores for entry into the study. The double-blind treatment phase will include a titration period of 3 weeks to determine the dosage, and a fixed-dosage period for the next 12 weeks. All patients who complete the double-blind treatment phase will be offered the option to enter the blinded extension phase for an additional 37 weeks, in which patients previously treated with carisbamate or placebo will receive carisbamate at their individual dosage at the end of the double-blind treatment period, and patients previously treated with pregabalin will receive pregabalin at their individual dosage at the end of the double-blind treatment period. During the double-blind and extension phases, patients will have daily assessments of their pain, using the 11-point DPN pain rating scale; and how much their pain interferes with their sleep, using an 11-point Sleep Interference rating scale. In addition, specific scales will be used at visits (every week for the first 4 weeks, every 4 weeks through the end of the double-blind treatment phase, every 11 to 12 weeks in the extension phase) to assess pain, overall health quality, the effects of pain on daytime sleepiness, and the effects of pain on work, activities, and health care utilization. Patients will remain blinded to the drug assignment during the extension phase. The posttreatment phase will include a follow-up visit with 7 to 14 days after the final visit of the double-blind treatment phase (for patients who do not participate in the extension phase) or the extension phase. In addition, the investigator staff will call patients 30 to 33 days after the last dose of study drug, to ask about any adverse events. Patients will take two oral capsules each day, either carisbamate (200 or 400 mg), matching pregabalin (75 or 150 mg), or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus (type 1 or 2)
* Have had diabetes-related painful peripheral neuropathy in the lower extremities for >=6 months prior to entry
* Have experienced lower extremity pain on a nearly daily basis for the previous 3 months
* Have a mean daily average DPN pain score of >=4 (on an 11-point scale) during the baseline period
* Have had a stable diabetic treatment regimen, including oral hypoglycemics, insulin, or diet, for >=3 months before screening
* Have hemoglobin A1c levels <=11%
* Willing to discontinue prohibited medications, including antiepileptic drugs (including gabapentin and pregabalin), opioids or opioid-containing pain medications, and antidepressants
* Women must be postmenopausal for >=2 years, surgically sterile, abstinent, or practicing a highly effective method of birth control
* Women of childbearing potential must have a negative pregnancy test at screening and on Day 1.

Exclusion Criteria:

* History of poor response to >=3 classes of medications for DPN
* Currently taking warfarin (Coumadin)
* Prior treatment with neurolysis (destruction of nerves by application of chemicals, heat, or cold), neurosurgery, intrathecal pumps, or spinal cord stimulators for DPN
* Use of herbal topical creams or ointments for pain relief with 48 hours, capsaicin with 6 months, or systemic (oral) corticosteroids with 3 months before the baseline period
* Any dermatologic or vascular disease in the limbs affected by the neuralgia that may interfere with assessment, including a diabetic ulcer or to or limb amputation
* Hospitalized within the last month for episodes of hypoglycemia or hyperglycemia
* History of progressive or neurologic disorders (such as multiple sclerosis, amyotrophic lateral sclerosis)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Mean of the last 7 daily average diabetic peripheral neuropathy (DPN) pain scores | Through 15 weeks

SECONDARY OUTCOMES:
Other secondary outcomes include the mean Neuropathic Pain Symptom Inventory (NPSI) subscale scores, the mean SF-36 subscale scores, and the Subject Global Impression of Change (SGIC) and Subject Global Impression of Severity (SGIS) scores. | Through 15 weeks
The proportion of patients who take rescue medication for breakthrough pain, and the number of days with rescue medication per week, will also be assessed. | Through 15 weeks
Responder rates (50% and 30% reduction from baseline in the mean of the last 7 daily average DPN pain scores). | Through 15 weeks
The mean of the last 7 daily maximum DPN pain scores. | Through 15 weeks
The mean of the last 7 Daily Sleep Interference scores. | Through 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.